CLINICAL TRIAL: NCT02914262
Title: Phase 1a Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of AKB 4924 in Healthy Male Volunteers
Brief Title: Single Ascending Dose Study to Assess the Safety, Tolerability, PK and PD Effects in Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerpio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AKB-4924-CI-1001
Record Dates: First submitted 2016-08-16; First posted 2016-09-26 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: IBD
MeSH Terms: interventions — AKB-4924

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental:Cohort 1-6 Experimental (Experimental): Intervention AKB 4924 Six subjects per cohort will receive single doses of 20 to up to 480 mg of AKB 4924 orally in a dose escalation format
  Interventions: Drug: AKB-4924
- Placebo:Cohort 1-6 (Placebo Comparator): Intervention Placebo:
  Two subjects per cohort will receive single oral doses of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AKB-4924 — Comparison of different dosages of AKB-4924
  Other Names: AKB-4924 Cohort 1-6
  Arms: Experimental:Cohort 1-6 Experimental
Other: Placebo — Placebo comparator
  Other Names: Placebo Cohort 1-5
  Arms: Placebo:Cohort 1-6

SUMMARY:
This will be a double-blind, randomized, placebo-controlled, single ascending dose, Phase I study in healthy male subjects.

DETAILED DESCRIPTION:
Single oral doses of AKB-4924 will be investigated in up to 6 sequential cohorts of 8 healthy male subjects. Primarily 6 dose levels are planned; the proposed doses are 20 mg, 60 mg, 120 mg, 240 mg, 360 mg, and 480 mg. Actual doses may be decreased or increased based on the safety and tolerability of the drug, as determined by the Investigator and Sponsor. Additional cohorts may be added as needed to test lower, higher, or repeat doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 to 49 years of age, inclusive.
2. Body mass index (BMI) between 18 to 30 kg/m2, inclusive.
3. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

1. Non-vasectomized male subjects and their female partners who are unable or unwilling to use an acceptable method of contraception (as described in Section 8.1.3, Contraception and Pregnancy Avoidance Measures) during the study and for 30 days following the last dose of study medication.
2. Evidence of active infection, unless the medical monitor and Investigator agree that the subject is appropriate for this study.
3. Current or past history of chronic disease including, but not limited to, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, neurologic, renal, or liver disease.
4. Diastolic blood pressure ≤55 mmHg or systolic blood pressure ≤100 mmHg at Screening.
5. Clinically important or significant conduction abnormalities on ECG at Screening (including QTcF intervals >450 msec) and/or history of long QT syndrome. It is acceptable to repeat the ECG to confirm findings.
6. Any history of malignancy in the previous 5 years except for curatively resected basal cell carcinoma of skin or squamous cell carcinoma of skin, or resected benign colonic polyps.
7. Seropositive for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibodies.
8. Serum transaminase (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) levels >1.5X the upper limit of normal (ULN). If a subject presents with an abnormal AST and/or ALT results, the subject may be re-scheduled or the test may be repeated once at the discretion of the Investigator.
9. Serum creatinine level ≥1.50 mg/dL. It is acceptable to repeat the test to confirm findings.
10. Chronic daily medication use, except once daily over the counter multi-vitamin supplement.
11. Subject has taken any prescription medication within 7 days (or 5 half-lives, whichever is longer) prior to admission to the CRU.
12. Herbal supplements within 48 hours prior to dosing of study drug.
13. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening.
14. Any history of alcohol or drug dependence within the previous year prior to Screening. Self-reported substance or alcohol dependence (excluding nicotine or caffeine) within the past 2 years, and/or have ever been in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence
15. Any use of alcohol within 48 hours of admission to the CRU.
16. Consumption of foods or beverages containing caffeine from 24 hours prior to dosing until the last sample collected during the Treatment period.
17. Subjects with a known history of smoking and/or has used nicotine or nicotine-containing products within the past 6 months.
18. Positive screen for drugs of abuse or a positive alcohol or cotinine result at screening or Day 1.
19. Donation of blood or blood products during the 4 weeks prior to dosing of study drug.
20. Physical activity greater than the normal level of activity from 48 hours prior to admission to the CRU.
21. Use of an investigational medication or device or participation in an investigational study within 30 days or 5 half-lives of the investigational medication, whichever is longer, preceding Day 1, or ongoing or scheduled participation in another investigational study during the present study through the Day 8 Follow-Up.
22. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the Investigator's judgment, would make the subject inappropriate for study entry.
23. Known allergy to HPβCD.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Single ascending dose (SAD): Safety and tolerability of AKB-4924 | 8 days after a single oral dose
  Safety evaluation will study the adverse event (AE) profile, clinical laboratory safety tests, vital signs and ECG monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonnell, MD, Principal Investigator — Syneos Health
Locations (1):
- INC Research, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No